CLINICAL TRIAL: NCT06616688
Title: Innovative Therapeutic Treatments to Inhibit Perineural Invasion in Pancreatic Adenocarcinoma
Acronym: PNIPDAC
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: National Nanotechnology Center (NANOTEC), The National Science and Technology Development Agency (NSTDA) (Unknown)
Responsible Party: Principal Investigator, Massimo Falconi, Head of Pancreatic Surgery, IRCCS San Raffaele
Other Study IDs: PNRR-MCNT1-2023-12378106
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Organoid-guided treatment — After specimen removal as per clinical practice and pathological examination, a small piece of tumor tissue will be sent to the Axo-Glial Interaction Unit and cultured to build up organoid cultures
  Other Names: Organoids colture

SUMMARY:
The overall goal of this project is to develop new therapeutic approaches to limit Perineural invasion (PNI) in pancreatic ductal adenocarcinoma (PDAC). PNI, has its higher incidence in PDAC, in which it is a recognized risk factor of poor survival. Considering the clinical relevance of PNI and its role in PDAC, it is urgent to identify molecular PNI signatures to develop new therapeutic strategies. We have recently identified a molecule that is activated in pancreatic cancer cells and initiate PNI. In this project we will hamper the signaling of this molecule in vitro, in human and murine organoids cocultured with myelinated Schwann cells neuronal cocultures, and in vivo in a mouse model faithfully reproducing human PNI. Thus, we will enroll patients undergoing surgical resection for PDAC, and a small piece of the resected tissue, performed for normal clinical practice after pathology evaluation, will be used to develop organoids.

This project is designed as an observational multicentric, transversal study. San Raffaele Hospital (OSR) is the only center enrolling patients.

The main goal of this Aim is to validate the effectiveness of NP-loaded hydrogel-based developed by CNR Nanotec Lecce, in vitro in organoids, which represent a suitable system to study PDAC.

DETAILED DESCRIPTION:
STUDY DESIGN The overarching goal of this project is to develop new therapeutic approaches to limit PNI formation and therefore PDAC formation and metastasis. PNI, has its higher incidence in PDAC, in which it is a recognized risk factor of poor survival. Considering the clinical relevance of PNI and its role in PDAC, it is urgent to identify molecular PNI signatures to develop new therapeutic strategies. We have recently identified a molecule (FGFBP1) that is activated in pancreatic cancer cells and initiate PNI.

This project is designed as an observational multicentric, cross-sectional study. OSR is the only center enrolling patients. OSR will send organoids derived from biological samples of enrolled patients to the participating center UO 3 (ASL3 Lecce) that will perform proteomic analyses to determine the level of expression of FGFBP1 inhibitor loaded in Nanoparticles hydrogels. Thus, the effectiveness of NP-loaded hydrogel carrying FGFBP1 inhibitors will be generated, and validated by CNR Nanotec Lecce (Aim 1, UO 2), whose biochemical release will be tested by mass spectrometry by UO 3 ASL3 Lecce; their biological effectiveness will be validated on myelinated Schwann cells neuronal cocultures seeded with human organoids carrying NP-loaded hydrogels (Aim 2 - OSR), and in vivo in TPAC mice, a recently developed animal model of PDAC, whose pancreas will be injected with NP-loaded hydrogels (Aim 3 - OSR).

Study duration Duration of enrollment: 18 months Duration of total follow-up: no follow-up needed for enrolled patients Duration of total study period: 24 months

STUDY POPULATION Study Participants Adult patients undergoing surgical pancreatic resection, as per clinical practice, with clinically and radiologically confirmed diagnosis of ductal adenocarcinoma. All patients will be enrolled at the OSR Pancreatic and Transplant Surgery Unit.

Inclusion Criteria

* Age 18 years (also fertile patients ca be included)
* Surgical resection for suspected PDAC, as per clinical practice. We will use this material both for controls and for the case samples.

Exclusion Criteria

* Patients who are not able to sign an informed consent
* Patients with suspected PDAC non confirmed at pathological report Screening Failures Participants who consented to participate in the clinical study, who do not meet one or more criteria required for participation in the study during the screening procedures, are considered screen failures.

STUDY OBJECT Study object description This is an observational study which does not require additional experimental procedures for the patients enrolled.

All patients will be treated according to guidelines regardless of their decision to participate in the study. All patients who do participate will sign the informed consent form attached to this protocol.

In Aim 1 (no human material required), UO 2 (CNR-Nanotech Lecce) will develop and characterize NP loaded hydrogels capable of releasing FGFBP1 inhibitors. Hydrogels will be characterized by rheometry, mechanical testing, morphological analysis, permeability/diffusion test, swelling and stability/degradation tests in physiological conditions. Cell studies (viability, morphology, motility, proliferation) will allow to evaluate the interaction between hydrogels and murine pancreatic cells to select the best performing compositions.

Obtained nanoparticles will be characterized: their surface charge, hydrodynamic diameter, particle distribution, and their stability in biological buffers will be monitored via light scattering technique. Nanoparticles' morphology will be studied using both scanning and transmission electron microscopy. FGFBP1 inhibitors loading, and release profiles under different stimuli will be monitored by advanced analytical techniques (chromatographic separations and detection by mass spectroscopy). Biocompatibility of the best nanoformulations will be assessed by performing viability assays, pro-inflammatory activities assays, cell cycle monitoring, hemolysis assay. These investigations will be carried out thanks to availability of instrumentation as flow cytometer, multimode plate reader and Laser Scanning Confocal Microscopy coupled with cell culture facility. Effective FGFBP1 inhibitor release will be tested by mass spectrometry analyses by UO 3 ASL3 Lecce using mass spectroscopy assays.

In Aim 2 UO 1 (OSR) will generate human and murine organoids from patients enrolled for surgical procedure after confirmed diagnosis of PDAC and from TPAC mice, respectively.

Organoids recapitulate the epithelial architecture of their organ of origin and reproduce the environmental signals present in both normal tissue and cancer while retaining the original genetic mutations.

Human pancreatic organoids will be prepared from PDAC patients whose diagnosis has been confirmed clinically and radiologically. Patients will be informed and asked to sign a consent for tissue collection. Resected specimens, collected in sterile conditions, will be transferred to the pathologist for a preliminary histological characterization. After isolating the tumor, the pathologist will provide us a small part of it that we will store in a 50 mL sterile tube in the presence of basal medium at 4°C for 16 hours to eliminate fat and blood cells. Next, we will separate cells from the surrounding fibrous tissue by mechanical dissection followed by enzymatic digestion with 0.125 mg/ml collagenase, 0.125 mg/ml dispase and 0.125 mg/ml DNAase. To remove the undigested material, we will pass it through a 40 μm cell strainer. All collected material will then be centrifuged, resuspend in cold Matrigel and plate in pre - warmed 4 well culture plates.

Murine organoids will be aldo prepared from the pancreas of TPAC mice, a recently developed animal model that develops PDAC and PNI from 12 months of age and faithfully reproduces the features of human cancer.

Both human and mouse collected tissue will be first mechanically dissociated and then enzymatically digested to obtain single cells. As control, we will either prepare naïve organoids and organoids embedded with hydrogels unloaded with FGFBP1 inhibitor. All cells will be resuspended in cold Matrigel and plated in pre-warmed 4 well culture plates.

Organoids will be also established from murine pancreas of the TPAC animal model characterized by extensive PNI in PDAC and from healthy murine pancreas, as control.

To validate the effectiveness of NP-loaded hydrogel-based, developed by UO 1 CNR Nanotec Lecce, in blocking FGFBP1 expression and limit PNI formation in PDAC, we will first perform proteomic analyses (UO 3 ASL3 Lecce) to monitor effective release of the inhibitor.

Effective inhibition of FGFBP1 will also be determined signaling in organoids loaded with FGFBP1 inhibitor hydrogels and relative controls by qRT-PCR (mRNA) and Western Blotting analyses (protein) by looking at specific downstream signaling effectors. The effect of hydrogels will be monitoed releasing FGFBP1 inhibitor onto organoids' growth and formation by scanning electron microscope and by immunofluorescence analyses for CK19, a marker of exocrine ductal cells and Sox 9, a marker of ductal lineage of pancreatic neoplasms. Schwann cells neuronal cocultureswill be established from E13.5 mouse dorsal root ganglia neurons as in (Taveggia and Bolino 2018), embed them in Matrigel to maintain comparable culture conditions with organoids, and let the cultures to myelinate for 21 days in the presence of 50 ug/ml ascorbic acid. Our preliminary data indicate that PDAC organoids seeded onto myelinated cocultures induce rapid and extensive myelin degeneration as assessed by MBP staining. Moreover, this event is rapidly blocked if PDAC organoids do not express FGFBP1. Thus, human and mouse organoids containing FGFBP1 inhibitor NP hydrogels and relative controls will be seeded, onto myelinated Schwann cells neuronal cocultures. The cultures will be manteined for additional 3, 7, 10, 15 and 21 days and monitor the extent of myelination and of axonal integrity by immunofluorescence analyses for MBP and NF.

Since in our preliminary data blocking FGFBP1 signaling rescues myelination, we expect that neuronal myelinated cocultures in contact with organoids loaded with NP hydrogels releasing FGFBP1 inhibitor will not degenerate unlike controls. Of particular interest, it will be to compare possible differences between human - and mouse-derived organoids.

In Aim 3 (no human material required), UO 1 will inject in the pancreas of TPAC mice, a recently developed animal model for PDAC, NP-loaded hydrogels releasing FGFB1 inhibitor.

The expression level of FGFBP1 will be first assesed at mRNA and protein level. and the expression of CK19 and Sox 9 (cancer cells), NF 200 (axons) and GFAP (SCs). All analyses will be done on 5 mice/group to reach statistical significance. In parallel, the expression levels of these protein will be also evaluated by Western Blotting analyses following standard protocols. To validate the effectiveness of NP-loaded hydrogels carrying FGFBP1 inhibitor, they will be inserted directly into the tail of the pancreas parenchyma of TPAC mice, by surgical procedures. In parallel, we hydrogels not containing nanoparticles will be injected in the pancreas of TPAC mice that will serve as negative controls. Tumor formation will be monitored by ultrasound analyses 10-, 20-, 30- 40- and 50-days post-hydrogel injection. Mice positive for tumor formation will undergo MRI analyses at the OSR Preclinical Imaging Facility to determine the presence of metastasis in close organs (liver / peritoneum). At the end of each time point, mice will be sacrificed, perfused in 4% PFA and the whole abdominal cavity included in OCT to analyze the histological characteristics of the primary tumor and assess the presence of PNI in the posterior nerve trunks and ganglia. 12 μm thick transverse sections will be cut at the cryostate, collected on Superfrost plus glass slides and processed for hematoxylin and eosin staining and immunofluorescence for CK 19, Sox 9 (cancer cells) and NF200 (axons). Spleen, duodenum, stomach, liver, kidneys, lungs, peritoneum and diaphragm will also be collected in 10% buffered formalin, embedded in paraffin wax and 3 μm sections stained with hematoxylin and eosin staining to detect metastasis formation.

SUBJECT RECRUITMENT AND SCREENING All surgically candidate patients for PDAC will be considered eligible for enrolling in the present study. The optimal goal would be to recruit at least 50 patients in the study period (18 months enrollment) A subject identification code will be assigned consecutively (i.e.: PNI_XXX; XXX is the progressive subject number in increasing order starting from 001).

A patient identification list will be kept. Baseline Assessments Baseline procedures coincide with the signing of informed consent for participation in the study. Being indeed a cross-sectional study no other procedures ad hoc for the study are planned for the participating patient.

SAMPLE HANDLING NP Loaded hydrogels releasing FGFBP1 inhibitors will be developed by UO 2 CNR Nanotec Lecce.

UO 1 will prepare human- and mouse-derived organoids carrying NP Loaded hydrogels releasing FGFBP1 inhibitors. UO 3, ASL3 Lecce, will determine effective release of FGFBP1 inhibitors in organoids by proteomic analyses.

Organoids will be established from surgically resected PDAC patients whose diagnosis of ductal adenocarcinoma was confirmed both clinically and radiologically at the OSR Pancreatic and Transplant Surgery Unit. Organoids will be established at the laboratory of Axo-Glial Interaction Unit (within OSR). All organoids of human and murine origin will be stored at the OSR CRB and in the laboratory of Axo-Glial interaction Unit at OSR for future studies, except part of and those carrying NP-loaded hydrogels that will be sent to the ASL3, Lecce, for proteomic analysis to validate effective release of the FGFBP1 inhibitor. After the analyses, which will last approximately 2 weeks, all organoids sent to ASL3 Leccesamples will return to OSR and destroyed.

Developed organoids carrying NP-loaded hydrogels will be validated in vitro onto Schwann cells neuronal myelinated cocultures for their effectiveness in limiting/blocking myelin degeneration. Preliminary data in fact indicate that blocking FGFBP1 activity blocks myelin degeneration in vitro and limit metastasis and PNI formation in vivo in mice.

NP-loaded hydrogels, upon validation, will also be implanted directly in the pancreas of TPAC mice, a recently developed model of PDAC. We will monitor tumor and PNI formation radiologically (ultrasound and MRI) and by histopathological analyses.

DATA MANAGEMENT Source Data: All information in original records and certified copies of original records of clinical findings, observations, or other activities in a clinical study necessary for the reconstruction and evaluation of the study. Source data are contained in source documents (original records or certified copies). Any data recorded directly on the CRFs (i.e., no prior written or electronic record of data), is considered to be source data.

Source Documents: Original documents, data, and records (e.g., hospital records; clinical and office charts; laboratory notes; memoranda) All parameters asked for in the case report form (CRF) will be documented in the source documents.

STATISTICS Description of Statistical Methods All generated data will be collected randomly (5 10X images collected at confocal microscope) and assessed blindly on samples of comparable size, especially for all in vitro analyses. Based on our experience we use a minimum of 5 biological replicates for each in vitro experiment. Thus, we will rely on the G-Power analyses to determine the minimum sample size required to obtain statically significant results with an impactful biological value.

Based on our previous comparable analyses, the data distribution will be assumed to be normal. All statistical analyses will be performed on at least five different experiments. Statistical detailed analyses will be assessed using Prism 9 Software package (GraphPad) and normally comprehend: Mann-Whitney test, ANOVA, with adjusted Bonferroni correction, Unpaired t test analyses, Ordinary OneWay Anova, Two-Way Anova, Tukey;s multiple comparison test.

All data generated during these procedures (such as optimization and characterization results obtained as function of the process parameters for hydrogel and nanoparticles preparation) will be collected and stored through dedicated repositories (e.g., Zenodo research data repository) and in data storage media (Dropbox Business).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years (also fertile patients ca be included)
* Surgical resection for suspected PDAC, as per clinical practice. We will use this material both for controls and for the case samples.

Exclusion Criteria:

* Patients < 18 years of age
* Patients who are not able to sign an informed consent
* Patients with suspected PDAC non confirmed at pathological report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing surgical pancreatic resection, as per clinical practice, with clinically and radiologically confirmed diagnosis of ductal adenocarcinoma. All patients will be enrolled at the OSR Pancreatic and Transplant Surgery Unit.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prepare and validate nanoparticles releasing FGFBP1 inhibitors | 8 months to assess hydrogels' safety and release of FGFBP1 inhibitors in NP-loaded hydrogels 12 months to complete the task
  Readout of these analyses will be the safety of developed hydrogels and effective release of FGFBP1 inhibitors.

SECONDARY OUTCOMES:
Treat peripheral myelinated cocultures with nanoparticles-loaded hydrogels targeting FGFBP1 signaling | Extent of myelin degeneration 3, 7-, 10-, 15- and 21-days post seeding human and mouse derived organoids mous
  Readout of these analyses will be the number of myelinated internodes (Myelin Basic Protein+ segments) in peripheral myelinated cocultures in the presence of organoids containing or not NP-loaded hydrogels.

IPD SHARING:
Plan to Share IPD: Yes
Required information will be valutated
Supporting Information: Study Protocol, SAP, CSR